CLINICAL TRIAL: NCT06324916
Title: Long Term Evaluation Of Donor Site Morbidities After Free Vascularized Fibular Graft For Reconstruction Of Any Bone Defect Other Than In The Lower Limb
Brief Title: Donor Site Morbidity After Free Vascularized Fibular Graft
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hedra Rafat Abdallah Ishak, Assistant Lecturer, Assiut University
Other Study IDs: vascularized fibular graft
Record Dates: First submitted 2023-09-21; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Xray — X rays for ankle to see distal fibular remenant

SUMMARY:
This study was carried out at Assiut University to Asses the long-term donor site morbidity following free vascularized fibular transfer because there is a limited information regarding the long-term donor morbidity of this type of flap.

DETAILED DESCRIPTION:
There is a dearth of information on the long-term donor site morbility of free fibular flaps. The recipient site can influence outcomes in the majority of research on donor site morbidity of free fibular grafting, but in this study, The invistigators will assess donor site morbidity and contrast the donor Leg with the contralateral Healthy one.

Surgical method for free fibular flapTo reduce ankle instability, the fibula was removed through lateral approach while the distal 5-7 cm of the bone was preserved. To seal the wound at the donor location, a full thickness or split thickness skin graft may be required. a suction drain that is implanted prior to healing. The donor leg was tightly covered with a bandage below the knee once the wound was closed. Using a skin graft to seal the wound.A gel foam pressure pack will be placed on top of an occlusive dressing if a skin transplant was utilized to seal the wound..

postoperative patients management: There was no difference in the postoperative care given to patients who had skin grafts at the donor location versus those who did not.

The entries in the patients' charts were used to evaluate postoperative wound healing at the donor site. It was determined whether wound healing was simple or involved. Dehiscence of wounds, necrosis of soft tissues,Patients will be questioned about when they first started using crutches and when they stopped using them after surgery, as well as when their ambulation returned to normal.

They were questioned about their subjective current symptoms of discomfort, pain, and edema, as well as about temperature differences, sensory abnormalities, motor function (i.e., range of motion), their ability to walk, run, ride a bike, and climb stairs, limitations on daily activities, and their satisfaction with the donor leg's scar's appearance.

During the physical examination in researchs, the donor leg was compared to the unoperated leg for the following parameters: strength and stability (ability to stand and walk on tiptoe and heels with both legs, with the unoperated and the operated leg); and sensory evaluation in specific areas of the calf. The latter included standardized examinations of pressure and touch perception (with a standardized pressure probe and cotton swab, respectively),the big toe was most frequently involved with weakness, both in flexion and extension. The muscle stripping of EHL and FHL during the harvest of the fibula is probably responsible for the weakness.

In this study,the invistigators will assess the outcomes and conduct data analysis to assess donor site morbidity and the benefits of surgery after free vascularized fibular transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients done FVFG for reconstruction of bone defect other than lower limb bone defect.
* surgery done >2yrs
* Patient age > 18 yrs old

Exclusion Criteria:

Patient age < 18 Surgery done< 2yrs FVFG for reconstruction of lower limb bone defct Amputated other leg : Above Ankle Amputaion Double FVFG Fracture of the other leg side : Fracture Tibia, Fibula, Ankle Paraplegic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a Retrospective Cohort study based on Assiut University microsurgery unit our target is All eligible patients during the period of the study will be included (total coverage sample).
  Expected number according to patients flow in the last year is 20 patients in Assiut University orthopedic surgery hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Donor site morbidity in contrast with surgery benifits this will be measured by point evaluation system | Two years after surgery
  in the point evaluation system patients filled out a questionnaire about the donor site scar, function loss, wound healing, complications, and pain. A total morbidity score was developed based on these items using a point rating system.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Taylor GI, Miller GD, Ham FJ. The free vascularized bone graft. A clinical extension of microvascular techniques. Plast Reconstr Surg. 1975 May;55(5):533-44. doi: 10.1097/00006534-197505000-00002. PMID 1096183
- [Background] Weinert CR Jr, McMaster JH, Ferguson RJ. Dynamic function of the human fibula. Am J Anat. 1973 Oct;138(2):145-9. doi: 10.1002/aja.1001380202. No abstract available. PMID 4747734
- [Background] Skraba JS, Greenwald AS. The role of the interosseous membrane on tibiofibular weightbearing. Foot Ankle. 1984 May-Jun;4(6):301-4. doi: 10.1177/107110078400400605. PMID 6735287
- [Background] Lee EH, Goh JC, Helm R, Pho RW. Donor site morbidity following resection of the fibula. J Bone Joint Surg Br. 1990 Jan;72(1):129-31. doi: 10.1302/0301-620X.72B1.2298771.
- [Background] Babhulkar SS, Pande KC, Babhulkar S. Ankle instability after fibular resection. J Bone Joint Surg Br. 1995 Mar;77(2):258-61. PMID 7706342
- [Background] Loro A, Hodges A, Galiwango GW, Loro F. Vascularized fibula flap in the management of segmental bone loss following osteomyelitis in children at a Ugandan hospital. J Bone Jt Infect. 2021 May 25;6(6):179-187. doi: 10.5194/jbji-6-179-2021. eCollection 2021. PMID 34109102
- [Background] Kanaya K, Wada T, Kura H, Yamashita T, Usui M, Ishii S. Valgus deformity of the ankle following harvesting of a vascularized fibular graft in children. J Reconstr Microsurg. 2002 Feb;18(2):91-6. doi: 10.1055/s-2002-19888. PMID 11823939
- [Background] Shingade VU, Jagtap SM, Ranade AB. Weakness of extensor hallucis longus after removal of non-vascularised fibula as an autograft. J Bone Joint Surg Br. 2004 Apr;86(3):384-7. doi: 10.1302/0301-620x.86b3.14748. PMID 15125126
- [Background] Di Giuli R, Zago M, Beltramini GA, Pallotta ML, Bolzoni A, Baj A, Gianni AB, Sforza C. Donor-Site Morbidity After Osteocutaneous Free Fibula Transfer: Longitudinal Analysis of Gait Performance. J Oral Maxillofac Surg. 2019 Mar;77(3):648-657. doi: 10.1016/j.joms.2018.10.016. Epub 2018 Nov 2. PMID 30481496
- [Background] Hakim SG, Tehrany AS, Wendlandt R, Jacobsen HC, Trenkle T, Sieg P. The impact of harvest length and detachment of the interosseous membrane on donor-site morbidity following free fibula flap surgery-a biomechanical experimental study. J Craniomaxillofac Surg. 2018 Nov;46(11):1939-1942. doi: 10.1016/j.jcms.2018.09.003. Epub 2018 Sep 19. PMID 30309796
- [Background] Zimmermann CE, Borner BI, Hasse A, Sieg P. Donor site morbidity after microvascular fibula transfer. Clin Oral Investig. 2001 Dec;5(4):214-9. doi: 10.1007/s00784-001-0140-5. PMID 11800433
- [Background] Hadouiri N, Feuvrier D, Pauchot J, Decavel P, Sagawa Y. Donor site morbidity after vascularized fibula free flap: gait analysis during prolonged walk conditions. Int J Oral Maxillofac Surg. 2018 Mar;47(3):309-315. doi: 10.1016/j.ijom.2017.10.006. PMID 29100670
- [Background] Goyal T, Paul S, Choudhury AK, Sethy SS. Full-thickness peroneus longus tendon autograft for anterior cruciate reconstruction in multi-ligament injury and revision cases: outcomes and donor site morbidity. Eur J Orthop Surg Traumatol. 2023 Jan;33(1):21-27. doi: 10.1007/s00590-021-03145-3. Epub 2021 Oct 26. PMID 34698925